CLINICAL TRIAL: NCT05326646
Title: Efficacy of a Low FODMAP Diet According to Colonic pH Measured by Wireless Motility Capsule in Irritable Bowel Syndrome Patients
Brief Title: Efficacy of a Low FODMAP Diet According to Colonic pH in Irritable Bowel Syndrome Patients
Acronym: FOSIIL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Medical Device (SmartPill) used in this project is no longer on the market
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019/0332/HP
Record Dates: First submitted 2021-12-08; First posted 2022-04-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: Low FODMAP diet; predictive factor; colonic pH
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBS patients (Experimental): Patients suffering from IBS according to Rome IV criteria
  Interventions: Dietary Supplement: Low FODMAP diet

INTERVENTIONS:
Dietary Supplement: Low FODMAP diet — After the realisation of a wireless motility capsule, patients will underwent 6 weeks of low FODMAP diet after dietician education. Symptomatic scores (IBS-SSS, GIQLI, HAD) and stools samples (metabolomic and lipidomic) will be performed before and after the low FODMAP diet.

SUMMARY:
Treatments efficacy in irritable bowel syndrome (IBS) patients is inconstant and predictive factors of their efficacy are needed. The role of dysbiosis in IBS is well-known. Another way to identify microbiota differences is to assess its metabolic activity. It has been demonstrated that colonic pH in IBS patients is lower than in healthy volunteers, reflecting a highest colonic fermentation. Colonic acidification is able to sensitize colonic mechano-receptors to distension. Microbiota profile is able to predict the response to a low Fermentable Oligo, Di, Monosaccharides And Polyols (FODMAPs) diet, but is not available in clinical routine.

The aim of our study is to assess the link between colonic fermentation (measured by colonic pH) and the efficacy of a low FODMAPs diet in IBS patients (measured by IBS severity scoring system (IBS-SSS)). We hypothesis that IBS patients with a lower colonic pH will have a better efficacy of the low FODMAPs diet. It might allow in the future personalized medicine.

50 IBS patients according to Rome IV criteria will be included in our study. All patients will have a measure of their colonic pH by wireless motility capsule. Patients will follow a low FODMAPs diet for 6 weeks after an education by a trained dietician. All participants will fill validated questionnaires before and after 6 weeks of low FODMAPs diet: IBS-SSS, Gastro Intestinal Quality of Life Index (GIQLI), Hospital Anxiety and Depression (HAD) scale. Microbiota, metabolomic and short chain fatty acid will be analysed before and after the intervention. The number of patients was calculated to assess the correlation between colonic pH and the variation of IBS-SSS before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* IBS according to Rome IV criteria
* Normal blood test (cell blood count, C Reactive Protein, thyroid-stimulating hormone, anti transglutaminase antibodies) in the last 12 months
* IBS severity score (IBS-SSS) >175/500
* IBS treatments stable in the last month
* Effective contraception since 1 month for women in childbearing age

Exclusion Criteria:

* Anorexia nervosa or any eating disorders deemed incompatible
* Organic gastroenterological diseases (inflammatory bowel disorder, microscopic colitis, gastrointestinal cancer, celiac disease)
* Contra-indication to the wireless motility capsule (intestinal stenosis, digestive fistula or obstruction, history of bezoar, gastrointestinal surgery in the last 3 months, acute diverticulitis, cardiac pacemaker, implanted electromedical device, magnetic resonance imaging planned in the 5 days after the wireless motility capsule, swallowing disorder)
* Breastfeeding or pregnant women
* Participation in another clinical trial in the last 2 weeks
* Patient who could not stop proton pump inhibitor treatment for 10 days
* Person with administrative or judicial decision or under legal protection measure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Correlation between efficacy of the low FODMAP diet on severity and the colonic pH | 6 weeks
  Correlation between colonic pH (baseline) and the variation of IBS severity score (IBS-SSS). IBS-SSS is a score between 0 (no symptom) to 500 (highest symptom level).

SECONDARY OUTCOMES:
Correlation between efficacy of the low FODMAP diet on quality of life and the colonic pH | 6 weeks
  Correlation between colonic pH (baseline) and variation of the quality of life Index (GIQLI). GIQLI is a score between 0 (lowest quality of life) and 144 (best quality of life).
Correlation between efficacy of the low FODMAP diet on stool frequency and the colonic pH | 6 weeks
  Correlation between colonic pH (baseline) and variation of the stool frequency
Correlation between efficacy of the low FODMAP diet on stool consistency and the colonic pH | 6 weeks
  Correlation between colonic pH (baseline) and variation of the stool consistency (BSF)
Correlation between efficacy of the low FODMAP diet on anxiety and the colonic pH | 6 weeks
  Correlation between colonic pH (baseline) and variation of anxiety (HAD). HAD anxiety is a scale comprised between 0 (no anxiety) and 21 (highest anxiety).
Correlation between efficacy of the low FODMAP diet on depression and the colonic pH | 6 weeks
  Correlation between colonic pH (baseline) and variation of depression (HAD). HAD depression is a scale comprised between 0 (no depression) and 21 (highest depression).
Correlation between short chain fatty acids and the colonic pH | 6 weeks
  Correlation between colonic pH (baseline) and variation of short chain fatty acids (in the stool)
Correlation between metabolites and the colonic pH | 6 weeks
  Correlation between colonic pH (baseline) and variation of metabolites (in the stool). Among metabolites, short chain fatty acids, 28 biliary acids and lipopeptides (C12-GABA, C12-Glutamine, C14-Glutamine, C15-GABA, C16-Glutamate, C16-Glutamine, C18-GABA, C12:1-Alanine (Ala)-GABA, C12-Ala-GABA, C13-Ala-GABA, C14:1-Ala-GABA et C183OH-Glutamate-GABA) will be assessed. Metabolites will be also assessed by RMN spectroscopy that allow the assessment of a high ranges of different metabolites.
Colonic pH according to small intestinal bacterial overgrowth | baseline
  Comparison of colonic pH between patients with and without small intestinal bacterial overgrowth
Colonic pH according to fructose malabsorption | baseline
  Comparison of colonic pH between patients with and without fructose malabsorption
Colonic pH according to visceral hypersensitivity | Baseline
  Comparison of colonic pH between patients with and without visceral hypersensitivity
Colonic pH and fecal calprotectin | Baseline
  Correlation between colonic pH and fecal calprotectin
Colonic pH and rectal pain threshold | Baseline
  Correlation between colonic pH and rectal pain threshold
Correlation between baseline QOL and the colonic pH | Baseline
  Correlation between colonic pH and baseline GIQLI (quality of life Index)
Correlation between baseline IBS severity score and colonic pH | Baseline
  Correlation between colonic pH and baseline IBS severity score (IBS-SSS)
Correlation between baseline anxiety and colonic pH | Baseline
  Correlation between colonic pH and baseline anxiety (HAD)
Correlation between baseline depression and colonic pH | Baseline
  Correlation between colonic pH and baseline depression (HAD)
Correlation between baseline stool consistency and colonic pH | Baseline
  Correlation between baseline stool consistency (BSF) and colonic pH
Correlation between baseline stool frequency and colonic pH | Baseline
  Correlation between baseline stool frequency and colonic pH

CONTACTS AND LOCATIONS:
Overall Officials: Chloé Melchior, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided
upon request